CLINICAL TRIAL: NCT02034760
Title: Counteracting Age-related Loss of Skeletal Muscle Mass
Acronym: CALM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Lars Holm, Ph.D. M.S., Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-4-2013-070
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Sarcopenia; Muscle Loss
Keywords: Frailty; Ageing; Protein supplementation; Protein quality; Gut microbiota; Metabolome; Exercise training; Sarcopenia
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Frailty | interventions — Whey; Carbohydrates

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Heavy Resistance Training (Active Comparator): Heavy Resistance Training of the lower extremities three times weekly in combination with two daily 20g whey protein and 10g carbohydrate supplementations for 52 weeks.
  Interventions: Procedure: Heavy Resistance Training; Dietary Supplement: Protein Whey
- Light Intensity Training (Experimental): Home-based Light Intensity Training of the lower extremities three-five times weekly in combination with two daily 20g whey protein and 10g carbohydrate supplementations for 52 weeks.
  Interventions: Procedure: Light Intensity Training; Dietary Supplement: Protein Whey
- Protein Whey (Active Comparator): Two daily 20g whey protein and 10g carbohydrate supplementations for 52 weeks.
  Interventions: Dietary Supplement: Protein Whey
- Protein Collagen (Active Comparator): Two daily 20g collagen protein and 10g carbohydrate supplementations for 52 weeks.
  Interventions: Dietary Supplement: Protein Collagen
- Carbohydrate (Placebo Comparator): Two daily 30g carbohydrate supplementations for 52 weeks.
  Interventions: Dietary Supplement: Carbohydrate

INTERVENTIONS:
Procedure: Heavy Resistance Training — Supervised Heavy Resistance Training three times weekly for 52 weeks.
  Arms: Heavy Resistance Training
Procedure: Light Intensity Training — Home-based Light Intensity Training three-five times weekly for 52 weeks.
  Arms: Light Intensity Training
Dietary Supplement: Protein Whey — Two daily 20g whey protein and 10g carbohydrate supplementations for 52 weeks.
  Arms: Heavy Resistance Training; Light Intensity Training; Protein Whey
Dietary Supplement: Protein Collagen — Two daily 20g collagen protein and 10g carbohydrate supplementations for 52 weeks.
  Arms: Protein Collagen
Dietary Supplement: Carbohydrate — Two daily 30g carbohydrate supplementations for 52 weeks.
  Arms: Carbohydrate

SUMMARY:
Up to approximately 205 (dependent on drop-out rate) healthy elderly individuals (at least 65 years old) are recruited as subjects.

Upon inclusion, each individual will be randomized into one of the five groups stratified according to gender (M/F) and 30s chair stand (<16 OR ≥16). The five groups are: Heavy Resistance Training (N=30-35), Light Intensity Training (N=30-35), Protein Whey (N=40-50), Protein Collagen (N=40-50) and Carbohydrate (N=30-35). The individuals randomized into one of the supplementation groups (Protein Whey, Protein Collagen or Carbohydrate) will be blinded to the supplement content.

Assessments will be performed at Baseline (before intervention start), and after 6 and 12 months of intervention and again at 18 months (after 6 months of follow up).

The primary outcome is change in quadriceps muscle cross sectional area from Baseline to 12 months of intervention.

The primary hypothesis is that by applying the intension-to-treat analysis, the Light Intensity Training group will increase quadriceps muscle cross sectional area just as much as the Heavy Resistance Training group. The two training groups will gain more muscle mass than the Protein Whey group, which will gain more than the Protein Collagen and the Carbohydrate groups that will loose quadriceps muscle cross sectional areas.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, independently living
* Age at least 65 years

Exclusion Criteria:

* Subjects dependent on help/nursing etc.
* Chronic medical diseases: Diabetes mellitus, clinical knee or hip osteoarthritis, other types of arthritis or connective tissue disorders, active cancer, renal diseases, severe chronic obstructive pulmonary disease, cardiac arrhythmias or known decreased left ventricular ejection fraction, lactose or gluten intolerance, chronic inflammatory bowel diseases, non-treated hyper/hypothyroidism, dementia.
* Surgical diseases: Bone, muscle, tendon or joint injuries compromising participation in exercise regimens.
* Implanted magnetic devices incompatible with MRi-scanning.
* Weekly alcohol consumption > 21 units (1 unit equals 4g of ethanol) for men and > 14 for women.
* Medicine except acetylsalicylic acid, paracetamol, thyroid function hormones, statins in doses above 40mg/day or if combined with subjective myalgia, ACE-inhibitors, Angiotensin II blockers, beta-blockers, calciumantagonists, proton-pump inhibitors, thiazides, potassium-sparing diuretics and loop diuretics.
* >1 hour of exercise weekly, except light activities such as stretching/gymnastics and bike-riding/walking as transportation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in muscle cross sectional area | Baseline, 6, 12, and 18 months
  MRi scans of quadriceps muscle cross sectional area. The primary time interval for assessment of the primary outcome measure is from Baseline to 12 months intervention. The statistical evaluation of the primary outcome measure is done by applying a two way ANOVA test comparing groups: 1) Heavy Resistance Training vs. Light Intensity Training vs. Protein Whey and 2) Protein Whey vs. Protein Collagen vs. Carbohydrate. The statistical evaluation will be performed first as an intension-to-treat analysis and subsequently as a per-protocol analysis.
  Assessments are performed at 6 months as well and at 18 months (after 6 months follow up). Changes in muscle cross sectional area will be evaluated over 6 months from Baseline to 6 months, from 6 to 12 months, and from 12 months to 18 months.

SECONDARY OUTCOMES:
Change in quadriceps muscle isometric strength | Baseline, 6, 12 and 18 months
  Isometric unilateral quadriceps force and rate of force development measured in the isokinetic dynamometer device (KinCom) during knee extension at the knee angle 70 deg (with 0 degrees being fully extended).
Change in quadriceps muscle isokinetic strength | Baseline, 6, 12 and 18 months
  Unilateral knee extension (concentric) strength measured in the KinCom device at an angular velocity of 60 degrees/sec.
Change in leg extension muscle power | Baseline, 6, 12 and 18 months
  Unilateral leg extension power measured in the Powerrig device.
Change from baseline in muscle structure and signalling | Baseline and 12 months
  From muscle biopsies muscle fiber type distribution and size, capillary density, satellite cell count and activity, selected gene-expression targets and protein concentrations will be assessed.
Change in gut microbiota composition. | Baseline, 6 and 12 months (and 18 months on a subset of samples).
  Molecular biology based methods incl. high throughput sequencing aided by classical, culture-based microbiological techniques as needed.
Change in faecal metabolome. | Baseline, 6 and 12 months (and 18 months on a subset of samples).
  NMR of faecal samples.
Change in faecal metabolome. | Baseline, 6 and 12 months (and 18 months on a subset of samples).
  Gas chromatography mass spectrometry (GCMS) of faecal samples.
Change in plasma metabolome. | Baseline, 6 and 12 months (and 18 months on a subset of samples).
  Nuclear magnetic resonance (NMR) of plasma samples.
Change in plasma metabolome. | Baseline, 6 and 12 months (and 18 months on a subset of samples).
  GCMS of plasma samples.
Change in 30 s chair stand | Baseline, 6, 12 and 18 months
  Number of stand-ups from a chair in 30 seconds.
Change in whole body composition and bone mineral density | Baseline, 6, 12 and 18 months
  Body composition (fat mass, lean mass and bone mass) evaluated by whole-body dual energy x-ray absorptiometry (DXA)-scanning.
  Bone mineral density at vertebrae L2-L4 and collum femoris evaluated by DXA-scanning.

OTHER OUTCOMES:
Change in blood parameters and anthropometry | Baseline, 6, 12 and 18 months
  Blood: HbA1c, plasma lipids, vitamin B12 and related metabolites. Anthropometry: Weight, abdominal circumference. Blood pressure.
Change in gait speed | Baseline, 6, 12 and 18 months
  400 m gait speed.
Change in grip strength | Baseline, 6, 12 and 18 months
  Isometric hand grip strength.
Change in tendon biomechanical properties | Baseline and 12 months
  Measurements of tendon biomechanical properties.
Questionnaires and interviews | Baseline and 12 months
  Short Form 36, Pittsburgh Sleep Scale Questionnaire, questionnaires on lifestyle, life history, supplement palatability and interviews and observations of subjects with focus on changes in lifestyle as result of intervention.
Change in daily macronutrient intake | Baseline, 1.5/2 and 12 months
  3-days self-report of food and beverage intake.
Change in habitual activity | Baseline, 6, 12 and 18 months
  Evaluated by 4 days continuous monitoring by a pedometer device (ActivPal).
Questionnaire on acceptance of supplements | Weekly for first 3 months and every 3rd month until 12 months
  Questionnaires on acceptance of supplementation
Change in glucose handling measured by a OGTT | Baseline and 12 months
  Completion of an oral glucose tolerance test (OGTT)
Change in vitamin B12 and related metabolite concentrations in blood | Baseline, 6, 12 and 18 months
  Concentration of total B12, B12 available for cells (holoTC), and methylmalonate (MMA).

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Bechshøft, Ph.d. stud, Principal Investigator — Bispebjerg Hospital; Lars Holm, Assoc. prof., Principal Investigator — Bispebjerg Hospital; Michael Kjaer, MD, Proff., Principal Investigator — Bispebjerg Hospital; Søren Reitelseder, Ph.d., Principal Investigator — Bispebjerg Hospital; Jacob Bülow, MD PhD stud, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispbebjerg Hospital, Copenhagen NV, Denmark

REFERENCES:
- [Derived] Mertz KH, Reitelseder S, Rasmussen MA, Bulow J, Hojfeldt G, Jensen M, Hjulmand M, Lindberg J, Kramer MU, Bechshoft R, Holm L. Changes in Muscle Mass and Strength During Follow-Up After One-Year Resistance Training Interventions in Older Adults. J Strength Cond Res. 2023 Oct 1;37(10):2064-2070. doi: 10.1519/JSC.0000000000004517. Epub 2023 Jul 17. PMID 37463344
- [Derived] Mertz KH, Reitelseder S, Bechshoeft R, Bulow J, Hojfeldt G, Jensen M, Schacht SR, Lind MV, Rasmussen MA, Mikkelsen UR, Tetens I, Engelsen SB, Nielsen DS, Jespersen AP, Holm L. The effect of daily protein supplementation, with or without resistance training for 1 year, on muscle size, strength, and function in healthy older adults: A randomized controlled trial. Am J Clin Nutr. 2021 Apr 6;113(4):790-800. doi: 10.1093/ajcn/nqaa372. PMID 33564844
- [Derived] Bechshoft RL, Reitelseder S, Hojfeldt G, Castro-Mejia JL, Khakimov B, Ahmad HF, Kjaer M, Engelsen SB, Johansen SM, Rasmussen MA, Lassen AJ, Jensen T, Beyer N, Serena A, Perez-Cueto FJ, Nielsen DS, Jespersen AP, Holm L. Counteracting Age-related Loss of Skeletal Muscle Mass: a clinical and ethnological trial on the role of protein supplementation and training load (CALM Intervention Study): study protocol for a randomized controlled trial. Trials. 2016 Aug 9;17(1):397. doi: 10.1186/s13063-016-1512-0. PMID 27507236